CLINICAL TRIAL: NCT01294969
Title: Patient Perception Study for AL-4943A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-10-15
Record Dates: First submitted 2011-02-10; First posted 2011-02-14 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2011-10

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AL-4943A (Experimental): One drop per day in both eyes
  Interventions: Drug: AL-4943A

INTERVENTIONS:
Drug: AL-4943A — Once daily topical ocular allergy medication used for 7 days

SUMMARY:
To evaluate patient perceptions of Al-4943 in subjects with allergic conjunctivitis previously treated with a topical ocular anti-allergy leukotriene-release inhibitor medication.

ELIGIBILITY:
Inclusion Criteria:

* History of allergic conjunctivitis within last 24 months
* Active signs and symptoms of ocular allergies

Exclusion Criteria:

* Severe or serious ocular condition, ocular surgical intervention, ocular infection

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Overall Patient satisfaction | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Korea Ltd., Seoul, South Korea